CLINICAL TRIAL: NCT03299283
Title: Specimen Collection and Transport Workflow Evaluations for CLIA-waived Molecular Testing
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: BioFire Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 804 Pilot
Record Dates: First submitted 2017-07-18; First posted 2017-10-03 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Respiratory Tract Infections; Gastrointestinal Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Respiratory and gastrointestinal specimens collected using medically established techniques
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Respiratory/Pharyngitis: Subject presents with signs/symptoms of respiratory infection including but not limited to fever, cough, sore throat (pharyngitis), runny nose, myalgia, headache, chills, or fatigue
  Interventions: Diagnostic Test: BioFire test platform
- Gastrointestinal: Subject presents with suspected gastroenteritis (e.g. diarrhea, vomiting, nausea, etc.) with duration of symptoms less than or equal to 7 days
  Interventions: Diagnostic Test: BioFire test platform

INTERVENTIONS:
Diagnostic Test: BioFire test platform — Analysis of analyte stability under various conditions as measured by BioFire test platforms

SUMMARY:
The purpose of this study is two-fold. In the first phase, the goal is to characterize the stability of respiratory (nasal swab, nasopharyngeal swab, and throat swab; NS, NPS, TS) and stool (raw stool and rectal swab) specimens collected using various standard, medically established procedures with and without transport media and tested at various time points and under different temperature conditions, and also to look at variation between repeat sampling events. The intention is for these data to support decisions made by BioFire regarding the appropriate specimen type and handling guidelines for future tests. In the second phase of the study, collection and transport conditions identified in Phase 1 will be used to collect specimens for pilot performance evaluations of a new molecular diagnostic test.

DETAILED DESCRIPTION:
This evaluation will be initiated at several sites in the US. In the first phase of the study, multiple specimens will be collected from each subject and tested using various pre-analytical techniques. Current BioFire FilmArray test panels will be used to assay each specimen and evaluate the multiple variables: repeat sampling, native specimen stability, or other post-collection variables. In the second phase of the study only two specimens will be collected from each subject: one for testing with the new test (using handling procedures identified in Phase 1) and another for testing with the reference method. Up to 2,000 subjects will be enrolled across all sites in each phase (up to 4,000 subjects total). Enrollment is expected to last approximately 18 months to cover both phases of the study. All specimens and subject data will be de-identified and coded. Prior to study initiation, each participating site will have the necessary Institutional Review Board (IRB) reviews. Specimens in both phases will be tested at the study site using various BioFire test platforms and cartridges.

ELIGIBILITY:
Inclusion Criteria:

* Subject presents with signs/symptoms of respiratory infection including but not limited to fever, cough, sore throat (pharyngitis), runny nose, myalgia, headache, chills, or fatigue. OR Subject presents with suspected gastroenteritis (e.g. diarrhea, vomiting, nausea, etc.) with duration of symptoms less than or equal to 7 days
* If age 18 or over, subject provides written informed consent
* If under the age of 18, parental permission and assent (as appropriate) is obtained
* Subject is willing and able to provide at least two (up to three) specimens: any combination of NS, NPS, or TS OR rectal swab or stool

Exclusion Criteria:

* Subject is unable to provide consent or parental permission and assent (as appropriate) cannot be obtained
* Subject is unable or unwilling to provide two specimens
* Subject's health care provider determines that specimen collection represents an unacceptable risk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects present to ED or urgent care centers with signs/symptoms of respiratory tract or gastrointestinal infection
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Analyte stability (as measured by nucleic acid detection) | Through completion of Phase 1 (approximartely 9 months)
  Sensitivity (or positive percent agreement) and specificity (or negative percent agreement) of the assays comprising the FilmArray Panel with respect to reference methods will investigate analyte stability for the various pre-analytical steps. Analyte stability will be measured by assessing nucleic acid level using real-time PCR.

SECONDARY OUTCOMES:
Device performance relative to reference methods | Through completion of Phase 2 (approximately 9 months)
  Sensitivity (or positive percent agreement) and specificity (or negative percent agreement) of the assays comprising the FilmArray Panel with respect to reference methods will determine device performance relative to reference method(s) i.e. if an anlyte is detected (or not) by each method (presence or absence)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Bourzac, PhD, Study Director — BioFire Diagnostics
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No